CLINICAL TRIAL: NCT06346470
Title: The Effect of Web-Based Breast Self-Examination Education on Nursing Students' Breast Self-Examination Knowledge, Skills, Attitude Towards Web-Based Instruction and Self-Directed Learning Skills: A Randomized Controlled Study
Brief Title: The Effect of Web-Based Breast Self-Examination Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, Dr, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3430-12
Record Dates: First submitted 2024-03-20; First posted 2024-04-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-03

CONDITIONS: Education; Breast Cancer
Keywords: breast cancer; breast self examination; web based education; nursing
MeSH Terms: conditions — Breast Neoplasms; Breast Self-Examination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web Based Breast Self-Examination Education Group (Experimental): For the web-based education group, a web page will be created by the researchers on Google classroom for breast self-examination skills. Prepared education materials will be uploaded to the website. Opinions of field experts will be sought for the prepared web page. The website will be rearranged in line with the suggestions of field experts. The education will last 6 hours in total.
  Interventions: Other: Web-based breast self examination education
- Traditional Breast Self-Examination Education Group (No Intervention): The group receiving education using the traditional method will be given breast self-examination education by the researchers. The education will cover topics such as the importance of breast self-examination, application times, and breast self-examination methods. Then, the breast self-examination skill will be taught using the technique of demonstrating and performing breast self-examination, and each student in the group will be allowed to perform the skill on the simulator. The education will last 4 hours in total.

INTERVENTIONS:
Other: Web-based breast self examination education — Students in this group will receive web-based breast self-examination education for 6 hours .
  Arms: Web Based Breast Self-Examination Education Group

SUMMARY:
Breast cancer is the most common type of cancer among women. Reasons such as diagnosing breast cancer at an early stage increases the chances of treatment and survival, and the fact that the masses are largely noticed by the individual themselves, point to the importance of breast self-examination (BSE) . BSE skill is among the nursing skills. When the literature was examined, it was seen that the web-based education method was frequently used for cognitive skills during nursing education, but its use was limited for psychomotor skills training. It was determined that in BSE training, in addition to traditional education, methods such as concept maps and peer-supported education were used, but web-based education methods were not used. It is thought that the study will contribute to the literature in these aspects.

DETAILED DESCRIPTION:
Due to the recent pandemic, nursing education, like other universities, was conducted web-based. Skills training in nursing, which is an applied education, has also been tried to be provided on a web-based basis. It is stated that the positive attitude towards e-learning increases the quality of education and student success. Additionally, with e-learning, the learner assumes individual learning responsibility. On the other hand, lack of motivation, attention, communication and interaction are the disadvantages of e-learning . Breast cancer is the most common type of cancer among women. Reasons such as diagnosing breast cancer at an early stage increases the chances of treatment and survival, and the fact that the masses are largely noticed by the individual themselves, point to the importance of breast self-examination (BSE). BSE skill is among the nursing skills. When the literature was examined, it was seen that the web-based education method was frequently used for cognitive skills during nursing education, but its use was limited for psychomotor skills training. It was determined that in BSE training, in addition to traditional education, methods such as concept maps and peer-supported education were used, but web-based education methods were not used. It is thought that the study will contribute to the literature in these aspects.

Hypotheses of the study;

H1: The BSE knowledge test score of the intervention group after the intervention is higher than the control group.

H2: BSE skill score of the intervention group is higher than the control group. H3: After the intervention, the intervention group's attitude towards web-based education is higher than the control group.

H4: After the intervention, the self-directed learning skills of the intervention group are higher than the control group.

H5: The initiative group's attitude towards web-based education increases after the initiative.

H6: Self-directed learning skills of the initiative group increase after the initiative.

ELIGIBILITY:
Inclusion Criteria:

- Being enrolled in the Surgical Nursing course (breast self-examination education is given for the first time within the scope of this course)

Exclusion Criteria:

- Having received breast self-examination education before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Skill and Knowledge of BSE | 2 weeks post intervention
  Skill and Knowledge of BSE point of the intervention group change after web based education
Attitude of Web-Based Education | 2 weeks post intervention
  Attitude of Web-Based Education point of the intervention group change after web based education
Self-Directed Learning Skills | 2 weeks post intervention
  Self-Directed Learning Skills point of the intervention group change after web based education

SECONDARY OUTCOMES:
Skill and Knowledge of BSE | 2 weeks post intervention
  The intervention group's BSE skill and knowledge score increased after the web-based training.
Self-Directed Learning Skills | 2 weeks post intervention
  Self-Directed Learning Skills point of the intervention group increased after web based education

CONTACTS AND LOCATIONS:
Overall Officials: Olga İncesu, PhD, Principal Investigator — İUC Florence Nightingale Faculty of Nursing
Locations (1):
- Florence Nightingale Faculty of Nursing, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No